CLINICAL TRIAL: NCT05082285
Title: A Phase II, Randomized, Partially Blinded Study to Assess the Safety, Tolerability and Immunogenicity of Meningococcal Combined ABCWY Vaccine When Administered to Healthy Infants
Brief Title: A Study on the Safety, Tolerability and Immune Response of Meningococcal Combined ABCWY Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217043; 2021-001367-24 (EudraCT Number)
Record Dates: First submitted 2021-10-07; First posted 2021-10-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Infections, Meningococcal
Keywords: MenABCWY-2Gen; MenABCWY-1Gen; Bexsero; Nimenrix; Safety; Tolerability; Immunogenicity; Invasive Meningococcal Disease; Healthy infants
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines; 4CMenB vaccine; tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ABCWY-2Gen low dose Group (Experimental): Participants receive 3 doses of the MenABCWY-2Gen low dose vaccine.
  Interventions: Combination Product: MenABCWY-2Gen low dose vaccine
- MenB+MenACWY-TT Group (Active Comparator): Participants receive 3 doses of both the meningococcal group B (MenB) vaccine and the meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate (MenACWY-TT) vaccine.
  Interventions: Combination Product: MenB vaccine; Combination Product: MenACWY-TT vaccine
- ABCWY-2Gen high dose Group (Experimental): Participants receive 3 doses of the MenABCWY-2Gen high dose vaccine in.
  Interventions: Combination Product: MenABCWY-2Gen high dose vaccine
- ABCWY-1Gen Group (Experimental): Participants receive 3 doses of the MenABCWY-1Gen vaccine.
  Interventions: Combination Product: MenABCWY-1Gen vaccine

INTERVENTIONS:
Combination Product: MenABCWY-2Gen low dose vaccine — MenABCWY-2Gen low dose vaccine is administered intramuscularly in the upper thigh region of the right leg as 3 doses to participants in study Part I, Step 1 and study Part II.
  Arms: ABCWY-2Gen low dose Group
Combination Product: MenABCWY-2Gen high dose vaccine — MenABCWY-2Gen high dose vaccine is administered intramuscularly in the upper thigh region of the right leg as 3 doses to participants in study Part I, Step 2 and study Part II.
  Arms: ABCWY-2Gen high dose Group
Combination Product: MenABCWY-1Gen vaccine — MenABCWY-1Gen vaccine is administered intramuscularly in the upper thigh region of the right leg as 3 doses to participants in study Part II.
  Arms: ABCWY-1Gen Group
Combination Product: MenB vaccine — MenB vaccine is administered intramuscularly in the upper thigh region of the right leg as 3 doses to participants in study Part I, Step 1 and Step 2 and study Part II.
  Other Names: Bexsero
  Arms: MenB+MenACWY-TT Group
Combination Product: MenACWY-TT vaccine — MenACWY-TT vaccine is administered intramuscularly in the lower thigh region of the right leg as 3 doses to participants in study Part I, Step 1 and Step 2 and study Part II.
  Other Names: Nimenrix
  Arms: MenB+MenACWY-TT Group

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of the combined meningococcal groups A, B, C, W and Y (MenABCWY-2Gen) vaccine intended to protect against invasive meningococcal disease (IMD) caused by all 5 meningococcal serogroups, in healthy infants 2 months of age (MoA) at enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 55 and 89 days of age (approximately 2 MoA) at the time of the first study vaccination.
* Born after a gestation period of ≥37 weeks, with a birth weight ≥2.5 kg.

Exclusion Criteria:

Medical conditions

* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection from birth.
* Progressive, unstable or uncontrolled clinical conditions.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any neuroinflammatory disorders, congenital and peripartum neurological conditions, encephalopathies, seizures.
* Congenital or peripartum disorders resulting in a chronic condition
* Major congenital defects, as assessed by the investigator.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s)/product(s).
* Hypersensitivity, including allergy, to any component of vaccines, including diphtheria toxoid (CRM197) and latex medicinal products or medical equipment whose use is foreseen in this study.
* Abnormal function or modification of the immune system resulting from:
* Autoimmune disorders or immunodeficiency syndromes.
* Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days starting from birth until Visit 5. This will mean prednisone equivalent ≥0.5 mg/kg/day with maximum 20 mg/day. Inhaled and topical steroids are allowed.
* Administration of antineoplastic and immunomodulating agents or radiotherapy from birth.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccines from birth, or planned use during the study period.
* Previous vaccination with any meningococcal vaccine.
* Administration of immunoglobulins and/or any blood products or plasma derivatives from birth or planned administration during the study period until Visit 5.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting from birth until Visit 5. For corticosteroids, this will mean prednisone equivalent ≥0.5 mg/kg/day with maximum 20 mg/day. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device).

Other exclusions

* Child in care.
* Study personnel as an immediate family or household member.
* For contraindications to administering routine vaccines foreseen in the study, refer to their approved product label/package insert.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 724 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with solicited administration site events | During the 7 days (including the day of vaccination) after each vaccination (vaccines administered on Day 1 and 61 and Day 301)
  The solicited administration site events include tenderness, erythema, induration and swelling.
Percentage of participants with solicited systemic events | During the 7 days (including the day of vaccination) after each vaccination (vaccines administered on Day 1 and 61 and Day 301)
  The solicited systemic events include fever, irritability/fussiness, loss of appetite, drowsiness, vomiting and diarrhoea. Fever is defined as temperature >38.0°C/100.4°F. The preferred location for measuring temperature will be axillary.
Percentage of participants with any unsolicited adverse events (AEs), including all medically attended adverse events (MAEs), serious adverse events (SAEs), AEs leading to withdrawal, and adverse events of special interest (AESIs) | During the 30 days (including the day of vaccination) after each vaccination (vaccines administered on Day 1 and 61 and Day 301)
  Unsolicited AEs includes any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. MAEs are defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it.
Percentages of participants with MAEs, SAEs, AEs leading to withdrawal, and AESIs | During the study period (Day 1 through Day 481)
  MAEs are defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it.
Percentage of participants with human serum bactericidal assay (hSBA) titers ≥ lower limit of quantitation (LLOQ) for each serogroup B indicator strain | At 1 month after the second vaccination (Day 91)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine is evaluated by measuring bactericidal activity using an hSBA against all serogroup B indicator strains.
Percentage of participants with hSBA titers ≥ LLOQ for each serogroup B indicator strain | At pre-third vaccination (Day 301)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine is evaluated by measuring bactericidal activity using an hSBA against all serogroup B indicator strains.
Percentage of participants with hSBA titers ≥ LLOQ for each serogroup B indicator strain | At 1 month after the third vaccination (Day 331)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine is evaluated by measuring bactericidal activity using an hSBA against all serogroup B indicator strains.
hSBA geometric mean titers (GMTs) for each serogroup B indicator strain | At 1 month after the second vaccination (Day 91)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine against serogroup B indicator strains is determined using hSBA GMTs. For each serogroup B indicator strain 90% CIs for the GMTs ratio between ABCWY-2Gen low dose/ ABCWY-2Gen high dose and MenB, is created by exponentiating (base 10) the least squares means and the lower and upper limits of the 90% CIs of the log transformed titers (base 10) obtained from a 2-way Analysis of Variance (ANOVA) with factors for arms and center.
hSBA GMTs for each serogroup B indicator strain | At pre-third vaccination (Day 301)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine against serogroup B indicator strains is determined using hSBA GMTs. For each serogroup B indicator strain 90% CIs for the GMTs ratio between ABCWY-2Gen low dose/ ABCWY-2Gen high dose and MenB, is created by exponentiating (base 10) the least squares means and the lower and upper limits of the 90% CIs of the log transformed titers (base 10) obtained from a 2-way ANOVA with factors for arms and center.
hSBA GMTs for each serogroup B indicator strain | At 1 month after the third vaccination (Day 331)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine against serogroup B indicator strains is determined using hSBA GMTs. For each serogroup B indicator strain 90% CIs for the GMTs ratio between ABCWY-2Gen low dose/ ABCWY-2Gen high dose and MenB, is created by exponentiating (base 10) the least squares means and the lower and upper limits of the 90% CIs of the log transformed titers (base 10) obtained from a 2-way ANOVA with factors for arms and center.
Within group hSBA geometric mean ratios (GMRs) for each serogroup B indicator strain | At 1 month after the third vaccination (Day 331) compared to pre-third vaccination (Day 301)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenB vaccine against serogroup B indicator strains is determined using hSBA GMRs. Within-group ratios of hSBA GMTs against each of the N.meningitidis serogroup B indicator strain at Day 331 compared to Day 301.
Percentage of participants with hSBA titers ≥ LLOQ for each A, C, W and Y serogroup | At 1 month after the second vaccination (Day 91)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine is evaluated by measuring bactericidal activity using an hSBA against serogroups A, C, W and Y. The percentages of participants with hSBA titers ≥ LLOQ and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method are calculated.
Percentage of participants with hSBA titers ≥ LLOQ for each A, C, W and Y serogroup | At pre-third vaccination (Day 301)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine is evaluated by measuring bactericidal activity using an hSBA against serogroups A, C, W and Y. The percentages of participants with hSBA titers ≥ LLOQ and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method are calculated.
Percentage of participants with hSBA titers ≥ LLOQ for each A, C, W and Y serogroup | At 1 month after the third vaccination (Day 331)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine is evaluated by measuring bactericidal activity using an hSBA against serogroups A, C, W and Y. The percentages of participants with hSBA titers ≥ LLOQ and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method are calculated.
hSBA GMTs for each A, C, W and Y serogroup | At 1 month after the second vaccination (Day 91)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine against serogroups A, C, W and Y is determined using hSBA GMTs. For each A, C, W, and Y serogroup 90% CIs for the GMTs ratio between ABCWY-2Gen low dose/ ABCWY-2Gen high dose and MenACWY-TT, is created by exponentiating (base 10) the least squares means and the lower and upper limits of the 90% CIs of the log transformed titers (base 10) obtained from a 2-way ANOVA with factors for arms and center.
hSBA GMTs for each A, C, W and Y serogroup | At pre-third vaccination (Day 301)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine against serogroups A, C, W and Y is determined using hSBA GMTs. For each A, C, W, and Y serogroup 90% CIs for the GMTs ratio between ABCWY-2Gen low dose/ ABCWY-2Gen high dose and MenACWY-TT, is created by exponentiating (base 10) the least squares means and the lower and upper limits of the 90% CIs of the log transformed titers (base 10) obtained from a 2-way ANOVA with factors for arms and center.
hSBA GMTs for each A, C, W and Y serogroup | At 1 month after the third vaccination (Day 331)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine against serogroups A, C, W and Y is determined using hSBA GMTs. For each A, C, W, and Y serogroup 90% CIs for the GMTs ratio between ABCWY-2Gen low dose/ ABCWY-2Gen high dose and MenACWY-TT, is created by exponentiating (base 10) the least squares means and the lower and upper limits of the 90% CIs of the log transformed titers (base 10) obtained from a 2-way ANOVA with factors for arms and center.
Within group hSBA GMRs for each A, C, W and Y serogroup | At 1 month after the third vaccination (Day 331) compared to pre-third vaccination (Day 301)
  The immune response to the MenABCWY-2Gen vaccine (low and high dose), the MenABCWY-1Gen vaccine and the MenACWY-TT vaccine against serogroups A, C, W and Y is determined using hSBA GMRs. Within-group ratios of hSBA GMTs against each of the N.meningitidis A, C, W and Y serogroups at Day 331 compared to Day 301.

CONTACTS AND LOCATIONS:
Locations (29):
- GSK Investigational Site, Santo Domingo Este, Dominican Republic
- Finland (6):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
- Germany (2):
  - GSK Investigational Site, Gilching
  - GSK Investigational Site, Schönau am Königssee
- GSK Investigational Site, San Pedro Sula, Honduras
- Poland (8):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Luboń
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- South Africa (2):
  - GSK Investigational Site, Parow Valley
  - GSK Investigational Site, Soweto Gauteng
- Spain (7):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- United Kingdom (2):
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.